CLINICAL TRIAL: NCT05242224
Title: Evolutionary Nutrition Pilot: Enhancing Fetal Growth and Brain Development
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Children's Discovery Institute (Other); Universidad San Francisco de Quito (Other); St. Louis Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-044E
Record Dates: First submitted 2019-06-28; First posted 2022-02-16 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Growth Disorders; Malnutrition, Fetal; Stunting; Development; Delayed, Malnutrition; Nutrition Disorder, Fetal; Maternal Nutritional Disorders Affecting Fetus or Newborn
MeSH Terms: conditions — Growth Disorders; Fetal Nutrition Disorders; Malnutrition

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Receives evolutionary nutrition package [high quality diet plus nutrition messaging + standard of care (iron-folic acid and calcium supplements)]
  Interventions: Other: Evolutionary Nutrition Package
- Control Group (No Intervention): Receives standard-of-care, iron-folic acid and calcium supplements.

INTERVENTIONS:
Other: Evolutionary Nutrition Package — The evolutionary nutrition package includes two key components: 1) one full meal per day from the evolutionary nutrition (EN) plate; 2) targeted messaging for high quality nutrition and removal of ultra-processed foods from the diet. The EN plate includes five food groups identified from the literature on evolutionary diets: animal source foods (ASF); berries and other fruits; tubers; vegetables, herbs and spices; and nuts and other legumes.
  Arms: Experimental Group

SUMMARY:
Globally, 250 million children do not reach their developmental potential and 155 million are stunted, yet few population-based studies have examined the direct effects of nutrient deficiencies on early brain development. This study will examine an evolutionary nutrition intervention during pregnancy derived from diets consumed for 99.9% of hominin history when bodies and brains were healthier. A pilot clinical trial will be conducted in the central highlands of Ecuador to compare fetal and newborn outcomes among women randomized to: 1) evolutionary nutrition package (high quality diet plus nutrition messaging); and 2) control (standard-of care supplements). Ultrasound brain measures, nutrition and morbidity data, and blood metabolomics will be assessed at 21 weeks gestational age, 37 weeks gestational stage, and postpartum. This pilot study uniquely combines the expertise of multiple disciplines - public health nutrition, radiology, neuroscience, and metabolomics - to examine the potential for improved nutrition on early growth and brain development with vital public health implications.

DETAILED DESCRIPTION:
The pilot trial will be conducted in the highlands of Ecuador in a mixed indigenous and non-indigenous population of pregnant women. Nationally, the stunting prevalence among young children is 25.3%, but large disparities within the country especially indigenous communities where stunting prevalence is nearly double, 42.3% (Freire et al., 2014). Incidence of low birthweight (8%) also varies by population in Ecuador, and may represent in utero growth restriction (IUGR) and other harmful exposures during pregnany (UNICEF 2012). While a large proportion of women have at least one antenatal care visit (84%), Only 58% of women in Ecuador meet the the WHO recommended 4+ antenatal care visits. This pilot project will leverage learnings from the Lulun Project and a previous antenatal health study (Gallegos et al. 2017) to design a social marketing campaign that encourages participation and high compliance. For this pilot RCT, the investigators will recruit pregnant women accessing antenatal care from Centro de Salud El Quinche in Pichincha province. Our target population will include those from poor households in particular (who access free public health services) with higher risks for IUGR and undernutrition during pregnancy.

The evolutionary nutrition package includes two key components: 1) one full meal per day from the evolutionary nutrition (EN) plate; 2) targeted messaging for high quality nutrition and removal of ultra-processed foods from the diet. The EN plate includes five food groups identified from the literature on evolutionary diets: animal source foods (ASF); berries and other fruits; tubers; vegetables, herbs and spices; and nuts and other legumes. In order to adapt the food groups to the Ecuador context, the investgators first developed a list of foods appropriate for the Ecuador context within each food group (Table 1). The food list draws on evidence from the Ministry of Health in Ecuador and USFQ for commonly consumed foods, notably among indigneous populations (Gallegos et al. 2010). Criteria for the full list of foods were the following: culturally appropriate; economically affordable and accessible; and environmentally sustainable. As was the experience with eggs in the Lulun Project, application of these criteria better ensure translation of findings within communities in the future.

Pregnant women will be recruited during first trimester of pregnancy and randomized to intervention group (EN plate + nutrition messaging + standard of care supplements) or control group (standard of care supplements). The intervention period will occur during second and third trimesters. Food supplies sufficient for one EN plate per day for 7 days will be delivered to pregnant women on a weekly basis. Under the supervision of the nutrition-trained field director, foods from each food group in pre-specified nutrient proportions will be secured from local food producers. Consideration will be given to including foods that do not require refrigeration over a one-week period. Careful documentation will be made of the foods contained in the weekly box in order to calculate exact quantity of nutrients provided. Due to concerns about food sharing that were evident in our qualitative research findings, additional food supplies will be provided for other household members in a separate container. Suggested menus and recipes will be provided with each delivery depending on the included foods.

Nutrition messages, developed in tandem with the social marketing campaign described below, will emphasize the importance of the food provisions for the participating pregnant women, but communicate the value of the EN plate for all household members. Messaging each week will reinforce the importance of eliminating ultraprocessed foods from the diet and reducing rice consumption. The absence of ultra processed foods is integral to our hypothesized effect and critical for confronting the dual burden of over- and under-nutrition in Ecuador (Freire et al. 2014). During each weekly food delivery visit, data will be collected on adherence and morbidities.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* in their first trimester
* carrying a singleton pregnancy

Exclusion Criteria:

* less than 18 years of age
* have a chronic health condition (HIV, TB, epilepsy, etc.)
* have a multiple pregnancy (twins, triplets, etc.)
* intend to move away from the study area
* have known allergies to eggs or fish
* have a blood pressure greater than 160/100

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-01-05 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Length-for-age Z (LAZ) | 6 months
  LAZ is a measure of stunting, whether a child is the appropriate length/height for their age
Plasma concentrations of Docosahexaenoic acid (DHA) | 6 months
  Plasma concentration of DHA measured in µg/mL
Plasma concentrations of Linoleic acid (LA) | 6 months
  Plasma concentration of LA measured in µg/mL
Plasma concentrations of α-Linoleic acid (ALA) | 6 months
  Plasma concentration of ALA measured in µg/mL
Plasma concentrations of Betaine | 6 months
  Plasma concentration of Betaine measured in µg/mL
Plasma concentrations of Methionine | 6 months
  Plasma concentration of Methionine measured in µg/mL
Plasma Concentration of Choline | 6 months
  Plasma concentration of Choline measured in µg/mL
Plasma Concentration of Iron (Fe) | 6 months
  Plasma concentration of Iron (Fe) measured in mg/mL
Plasma Concentration of Zinc (Zn) | 6 months
  Plasma concentration of Zinc (Zn) measured in mg/mL
Plasma Concentration of Selenium (Se) | 6 months
  Plasma concentration of Selenium (Se) measured in mg/mL
Brain structure development--Gangliothalamic ovoid (GTO) volume | 4 months
  GTO volume measured in cm3
Brain structure development--Gangliothalamic ovoid (GTO) diameter | 4 months
  GTO diameter measured in cm
Brain structure development--Gangliothalamic ovoid (GTO) craniocaudal | 4 months
  GTO craniocaudal measured in cm
Brain structure development-- thalamic diameter | 4 months
  Thalamic diameter in cm

SECONDARY OUTCOMES:
Maternal Morbidity | 6 months
  Rate of morbidities common during pregnancy including anemia, urinary tract infections, hypertension, gestational diabetes, respiratory infections, and hyperemesis gravidarum.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Palacios, MD, Study Director — Universidad San Francisco de Quito
Locations (1):
- Universidad San Francisco de Quito, Quito, Pichincha, Ecuador